CLINICAL TRIAL: NCT07158606
Title: Understanding Treatment Outcomes and Immunologic Mechanisms in ALtuviiio Immune Tolerance Induction
Acronym: UTILITI
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Versiti Blood Health (Other)
Responsible Party: Principal Investigator, Lynn Malec, Medical Director, Versiti Comprehensive Center for Bleeding Disorders, Versiti Blood Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00052811
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A With Inhibitor
MeSH Terms: interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ITI (Experimental): ITI therapy will involve subjects receiving efanesoctacog alpha at a determined dose.
  Interventions: Drug: efanesoctacog alpha; Drug: Emicizumab

INTERVENTIONS:
Drug: efanesoctacog alpha — Efanesoctacog alpha will be administered at a dose of 50 IU/kg two times weekly during the ITI Treatment Period. The site investigator will determine the dose of efanesoctacog alpha once the subjects reaches the Follow Up Period.
Drug: Emicizumab — Emicizumab will be prescribed as standard of care bleed prevention.

SUMMARY:
The goal of this clinical trial is to learn how well Altuviiio (efanesoctacog alpha) works for Immune Tolerance Induction (ITI) while using Hemlibra (emicizumab) to prevent bleeds.

Participants will be given Altuviiio for their ITI therapy and also be treated with Hemlibra as standard of care prophylaxis to prevent bleeding. The research doctor will decide how much and how often the participant will get Hemlibra.

Participants will need to attend visits for checkups and tests. These visits are divided into 4 periods:

1. A screening period - 1 visit up to 8 weeks before the Treatment Period starts
2. ITI Treatment Period - 1 Baseline Visit plus Interim visits that occur every 4 weeks for up to 52 weeks. (Some of the interim visits may be done via phone)
3. Tapering Period - 5 visits at weeks 2, 4, 8, 12 and 16
4. Ongoing Monitoring Period - 4 visits at weeks 20, 30, 40 and 50

ELIGIBILITY:
Inclusion Criteria:

1) severe hemophilia A (congenital) 2) history of high titer inhibitor (≥ 5 BU) 3) peak inhibitor titer (pre-ITI) < 1,000 3) age < 18 y/o at the time of study enrollment 4) undergoing initial ITI course 5) current or planned concomitant use of emicizumab

Exclusion Criteria:

1. von Willebrand disease or a known second bleeding diathesis besides SHA
2. prior course of ITI
3. inhibitor present for > 2 years without prior attempts at eradication

3) personal history of unprovoked thrombosis 4) known contraindication, intolerance, or allergy to either of the investigational agents of study 5) inability or unwillingness to provide informed consent and/or assent 6) inability to speak or read English 7) Any other condition, that in the opinion of the investigator, would negatively impact the safety of the participant

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
ITI Success | 12 months
  Time from initial dose of efanesoctacog alpha for ITI to ITI success or failure.

SECONDARY OUTCOMES:
Events | 12 months
  All bleeding events and factor and bypassing agent consumption from the time of ITI initiation until a patient has achieved tolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Versiti Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided